CLINICAL TRIAL: NCT02733016
Title: Seinäjoki Adult Asthma Study: A 12-year Real-life Follow-up Study of New-onset Asthma Diagnosed at Adult Age and Treated in Primary and Specialized Care. Finnish Title: Diagnoosista Hoitotasapainoon: Voidaanko Aikuisen Astman Hoitotasapainoa Ennustaa Diagnoosivaiheen löydösten ja Astman Ilmiasun Perusteella?
Brief Title: Seinäjoki Adult Asthma Study
Acronym: SAAS
Status: Completed | Type: Observational
Sponsor: Seinajoki Central Hospital (Other)
Responsible Party: Principal Investigator, Hannu Kankaanranta, Professor and Head of Respiratory Medicine, Seinajoki Central Hospital
Other Study IDs: SCH-2000
Record Dates: First submitted 2016-03-16; First posted 2016-04-11 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Seinäjoki Adult Asthma Study is a single-centre 12-year follow-up study of a total cohort of 259 patients having new-onset asthma that was diagnosed at adult age. The study was divided in two parts: the collection of the original cohort (phase I;n=259) and follow-up visit (phase II; n=203). The aim of this study is to increase the understanding on the diagnostics and diagnostic process, organisation of the long-term asthma care, therapeutic outcomes, prognosis and the factors affecting the prognosis of new-onset asthma diagnosed at adult age.

DETAILED DESCRIPTION:
At baseline visit the diagnostic studies performed were: spirometry, PEF (peak expiratory flow) follow-up, other respiratory physiology measurements, laboratory, skin-prick, AQ20 (Airways questionnaire 20), 15D, background data. At follow-up visit, asthma status, co-morbidities (chronic rhinitis or obstructed nose, allergic rhinitis or conjunctivitis, diabetes, hypertension, coronary heart disease, COPD (chronic obstructive pulmonary disease) and any other patient-reported disease), medication (including medication to other diseases and the disease treated), control, severity and lung function were evaluated. In addition to the data gathered at these visits, data on asthma follow-up visits, exacerbations, hospitalisations, possible occupationally induced asthma and prescribed asthma medication were collected from hospital clinics, primary health care, occupational health care and private practices for the whole 12-year follow-up period. In addition, the use of medication that was realised, i.e., medication bought from pharmacy, will be retrieved. In addition to asthma-specific factors, data include occupational, lifestyle and socioeconomic factors at the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of new-onset asthma made by a respiratory specialist
* Diagnosis confirmed by at least one of the following objective lung function measurements

  * FEV1 (forced expiratory volume in one second) reversibility in spirometry of at least 15% and 200 ml
  * Diurnal variability (⩾20%) or repeated reversibility (⩾15%/60 l/min) in PEF follow-up
  * A significant decrease in FEV1 (15%) or PEF (20%) in response to exercise or allergen
  * A significant reversibility in FEV1 (at least 15% and 200 ml) or significant mean PEF in response to a trial with oral or inhaled glucocorticoids
  * Symptoms of asthma
  * Age ≥15 years

Exclusion Criteria:

* Physical or mental inability to provide signed informed consent
* Diagnosis of asthma below the age of 15 years

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort of 259 patients having new-onset asthma that was diagnosed at adult age. Patients were referred to the hospital by primary-care practitioners because of suspicion of asthma. After 12 years, patients were invited to a follow-up visit. Total of 203 patients returned to follow-up visit.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 1999-10; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Asthma control at follow-up visit | 12 years
  Asthma control at follow-up visit according to GINA (Global Initiative for asthma) report 2010.

SECONDARY OUTCOMES:
Remission of asthma at follow-up visit | 12 years
  Four different criteria for remission are defined:1) no reported symptoms of asthma in the structured questionnaire, 2) Asthma Control Test (ACT) score of 25, 3) no use of medication for asthma during last 6 months, and 4) no use of oral prednisolone courses during the last 2 years. Further definitions included also normal lung function.
Annual number of asthma exacerbations during follow-up period | 12 years
  Exacerbations as defined by number of prescriptions of oral steroid courses due to asthma, during the follow-up period.
Annual number of asthma-related visits to healthcare | 12 years
  All asthma-related visits to healthcare during the follow-up period are recorded.
Annual number of asthma control visits | 12 years
  All asthma control visits (primary care, specialized care, occupational health care, private health care) during the follow-up period are recorded.
Annual asthma-related hospitalizations | 12 years
  All asthma-related hospitalizations during the whole follow-up period are recorded.
Proportion of asthma control visits performed at primary health care | 12 years
  Proportion of asthma control visits performed at primary health care (either physician or nurse)
Proportion of diagnoses of asthma that are based on spirometry | Diagnosis
  Proportion of diagnoses that are solely based on spirometry (FEV1 reversibility of at least 15 % and 200 ml or reversibility in response to a trial with oral or inhaled corticosteroids or a significant decrease in FEV1 (15 %) in response to exercise or allergen).
Proportion of diagnoses of asthma that are based on PEF (Peak Expiratory Flow) | Diagnosis
  Proportion of diagnoses that are solely based on PEF measurement (diurnal variability (≥ 20 %) or repeated reversibility (≥ 15 % / 60 L / min) in PEF-follow-up or significant mean PEF in response to a trial with oral or inhaled glucocorticoids or a significant decrease in PEF (20 %) in response to exercise or allergen).
Blood eosinophils at diagnostic and follow-up visits | 12 years
  Venous blood is collected and white blood cells including eosinophils counted
Blood neutrophils at follow-up visit | 12 years
  Venous blood is collected and white blood cells including neutrophils counted
Fraction of expiratory nitric oxide (FeNO) at follow-up visit | 12 years
  Fraction of exhaled nitric oxide (FENO) is measured with a portable rapid-response chemiluminescent analyzer according to ATS (American Thoracic Society) standards
Airways questionnaire 20 (AQ20) score at diagnostic and follow-up visit | 12 years
  AQ20 is a validated tool to evaluate symptoms of asthma and asthma-related quality of life.
Asthma control test (ACT) score at follow-up visit | 12 years
  Asthma control test is a validated tool, an international structured questionnaire to evaluate symptoms and control of asthma.
Total Immunoglobulin E (IgE) at diagnosis and follow-up | 12 years
  Total IgE levels as measured by using ImmunoCAP.
Annual change in FEV1 during follow-up | 1 year
  Annual change in FEV1 from point of maximal lung function within 2.5 yrs after diagnosis (and start of therapy) to follow-up visit
Proportion of daily users of inhaled steroids at follow-up visit | 12 years
  Use of inhaled steroids is evaluated based on a structured questionnaire.
Proportion of users of daily add-on medication at follow-up visit | 12 years
  Use of add-on medication (long-acting beeta2-agonists, leukotriene receptor antagonists, tiotropium or theophylline) is evaluated based on a structured questionnaire.
Leptin at follow-up visit | 12 years
  Leptin was measured by ELISA at follow-up visit.
Adiponectin at follow-up visit | 12 years
  Adiponectin was measured by ELISA at follow-up visit.
YKL-40 at follow-up visit | 12 years
  YKL-40 was measured by ELISA at follow-up visit.
Pre-bronchodilator FEV1 at follow-up visit | 12 years
  Spirometry was performed according to international recommendations.
Post-bronchodilator FEV1 at follow-up visit | 12 years
  Spirometry was performed according to international recommendations.
Pre-bronchodilator FEV1/FVC (Forced Vital Capacity) at follow-up visit | 12 years
  Spirometry was performed according to international recommendations.
Post-bronchodilator FEV1/FVC at follow-up visit | 12 years
  Spirometry was performed according to international recommendations.
Pre-bronchodilator FVC (Forced Vital Capacity) at follow-up visit | 12 years
  Spirometry was performed according to international recommendations.
Post-bronchodilator FVC at follow-up visit | 12 years
  Spirometry was performed according to international recommendations.
Proportion of patients with asthma-COPD overlap syndrome at follow-up visit | 12 years
  Proportion of patients fulfilling also criteria of COPD: at least 10 smoked pack years and post-FEV1/FVC<0,7.
Rhinitis at follow-up | 12 years
  Allergic or non-allergic rhinitis or persistent rhinitis as evaluated by structured questionnaire.
high sensitivity C-reactive protein (hsCRP) concentration at follow-up | 12 years
  hsCRP is measured using particle-enhanced immunoturbidometric method.
serum interleukin-6 (IL-6) at follow-up | 12 years
  serum levels of IL-6 are measured by ELISA assay.
Quality of life index 15D at baseline and at follow-up | 12 years
  15D is a validated tool to measure quality of life
Number of co-morbidities at follow-up visit | 12 years
  Number and quality of co-morbidities at follow-up visit will be evaluated by using structured questionnaire and from patients records
Number of other medications | 12 years
  Number of other medications at follow-up visit will be evaluated by structured questionnaire
Number or current and ex-smokers and smoked pack-years at baseline and follow-up | 12 years
  Number or current and ex-smokers and smoked pack-years at baseline and follow-up will be evaluated by using structured questionnaire
BMI (body-mass index) at baseline and follow-up and BMI change during follow-up | 12 years
  Weight, height were collected at baseline and at follow-up and BMI calculated
Proportion of patients using at least 2 oral steroid bursts during last 2 years | 2 years
  Proportion of patients having used at least 2 oral steroid bursts during last 2 years evaluated by using structured questionnaire
Use of alcohol and coffee at follow-up | 12 years
  Use of alcohol and coffee at follow-up evaluated by using structured questionnaire
Daily time spent sitting at follow-up | 12 years
  Daily time spent in sitting position at follow-up evaluated by structured questionnaire
Weekly exercise frequency at follow-up | 12 years
  Weekly exercise frequency at follow-up evaluated by structured questionnaire
Daily screen time at follow-up | 12 years
  Daily time spent in front of the screen evaluated at follow-up by structured questionnaire
Glutamyl transferase at follow-up | 12 years
  Glutamyl transferase at follow-up evaluated by routine standard laboratory methods
Carbohydrate-deficient transferrin (CDT) at follow-up | 12 years
  CDT at follow-up measured by using routine standard laboratory methodology

CONTACTS AND LOCATIONS:
Overall Officials: Hannu Kankaanranta, Professor, Principal Investigator — Seinajoki Central Hospital
Locations (1):
- Department of Respiratory Medicine, Seinäjoki Central Hospital, Seinäjoki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kankaanranta H, Ilmarinen P, Kankaanranta T, Tuomisto LE. Seinajoki Adult Asthma Study (SAAS): a protocol for a 12-year real-life follow-up study of new-onset asthma diagnosed at adult age and treated in primary and specialised care. NPJ Prim Care Respir Med. 2015 Jun 25;25:15042. doi: 10.1038/npjpcrm.2015.42. No abstract available. PMID 26110580
- [Background] Ilmarinen P, Tuomisto LE, Kankaanranta H. Phenotypes, Risk Factors, and Mechanisms of Adult-Onset Asthma. Mediators Inflamm. 2015;2015:514868. doi: 10.1155/2015/514868. Epub 2015 Oct 11. PMID 26538828
- [Background] Tuomisto LE, Ilmarinen P, Kankaanranta H. Prognosis of new-onset asthma diagnosed at adult age. Respir Med. 2015 Aug;109(8):944-54. doi: 10.1016/j.rmed.2015.05.001. Epub 2015 May 21. PMID 26052036
- [Background] Kankaanranta H, Kauppi P, Tuomisto LE, Ilmarinen P. Emerging Comorbidities in Adult Asthma: Risks, Clinical Associations, and Mechanisms. Mediators Inflamm. 2016;2016:3690628. doi: 10.1155/2016/3690628. Epub 2016 Apr 26. PMID 27212806
- [Background] Kankaanranta H, Tuomisto LE, Ilmarinen P. Age-specific incidence of new asthma diagnoses in Finland. J Allergy Clin Immunol Pract. 2017 Jan-Feb;5(1):189-191.e3. doi: 10.1016/j.jaip.2016.08.015. Epub 2016 Oct 17. No abstract available. PMID 27765463
- [Result] Tuomisto LE, Ilmarinen P, Niemela O, Haanpaa J, Kankaanranta T, Kankaanranta H. A 12-year prognosis of adult-onset asthma: Seinajoki Adult Asthma Study. Respir Med. 2016 Aug;117:223-9. doi: 10.1016/j.rmed.2016.06.017. Epub 2016 Jun 23. PMID 27492535
- [Result] Ilmarinen P, Tuomisto LE, Niemela O, Danielsson J, Haanpaa J, Kankaanranta T, Kankaanranta H. Comorbidities and elevated IL-6 associate with negative outcome in adult-onset asthma. Eur Respir J. 2016 Oct;48(4):1052-1062. doi: 10.1183/13993003.02198-2015. Epub 2016 Aug 18. PMID 27540019
- [Result] Tommola M, Ilmarinen P, Tuomisto LE, Haanpaa J, Kankaanranta T, Niemela O, Kankaanranta H. The effect of smoking on lung function: a clinical study of adult-onset asthma. Eur Respir J. 2016 Nov;48(5):1298-1306. doi: 10.1183/13993003.00850-2016. Epub 2016 Sep 22. PMID 27660515
- [Result] Ilmarinen P, Tuomisto LE, Niemela O, Tommola M, Haanpaa J, Kankaanranta H. Cluster Analysis on Longitudinal Data of Patients with Adult-Onset Asthma. J Allergy Clin Immunol Pract. 2017 Jul-Aug;5(4):967-978.e3. doi: 10.1016/j.jaip.2017.01.027. Epub 2017 Apr 25. PMID 28389304
- [Result] Tommola M, Ilmarinen P, Tuomisto LE, Lehtimaki L, Haanpaa J, Niemela O, Kankaanranta H. Differences between asthma-COPD overlap syndrome and adult-onset asthma. Eur Respir J. 2017 May 1;49(5):1602383. doi: 10.1183/13993003.02383-2016. Print 2017 May. PMID 28461298
- [Result] Tommola M, Ilmarinen P, Tuomisto LE, Kankaanranta H. Concern of underdiagnosing asthma-COPD overlap syndrome if age limit of 40 years for asthma is used. Eur Respir J. 2017 Aug 3;50(2):1700871. doi: 10.1183/13993003.00871-2017. Print 2017 Aug. No abstract available. PMID 28775049
- [Result] Vahatalo I, Ilmarinen P, Tuomisto LE, Niemela O, Kankaanranta H. Inhaled corticosteroids and asthma control in adult-onset asthma: 12-year follow-up study. Respir Med. 2018 Apr;137:70-76. doi: 10.1016/j.rmed.2018.02.025. Epub 2018 Mar 2. PMID 29605216
- [Result] Ilmarinen P, Tuomisto LE, Niemela O, Kankaanranta H. Prevalence of Patients Eligible for Anti-IL-5 Treatment in a Cohort of Adult-Onset Asthma. J Allergy Clin Immunol Pract. 2019 Jan;7(1):165-174.e4. doi: 10.1016/j.jaip.2018.05.032. Epub 2018 Jun 9. PMID 29894793
- [Derived] Nordman L, Vahatalo I, Tuomisto LE, Niemela O, Tommola M, Lehtimaki L, Ilmarinen P, Kankaanranta H. Risk factors for asthma exacerbations. J Allergy Clin Immunol Glob. 2025 Jun 21;4(3):100520. doi: 10.1016/j.jacig.2025.100520. eCollection 2025 Aug. PMID 40697950
- [Derived] Takala J, Vahatalo I, Tuomisto LE, Niemela O, Ilmarinen P, Kankaanranta H. Participation in scheduled asthma follow-up contacts and adherence to treatment during 12-year follow-up in patients with adult-onset asthma. BMC Pulm Med. 2022 Feb 15;22(1):63. doi: 10.1186/s12890-022-01850-1. PMID 35168565
- [Derived] Ilmarinen P, Vahatalo I, Tuomisto LE, Niemela O, Kankaanranta H. Long-term adherence to inhaled corticosteroids in clinical phenotypes of adult-onset asthma. J Allergy Clin Immunol Pract. 2021 Sep;9(9):3503-3505.e3. doi: 10.1016/j.jaip.2021.04.057. Epub 2021 May 30. No abstract available. PMID 33965594
- [Derived] Ilmarinen P, Pardo A, Tuomisto LE, Vahatalo I, Niemela O, Nieminen P, Kankaanranta H. Long-term prognosis of new adult-onset asthma in obese patients. Eur Respir J. 2021 Apr 1;57(4):2001209. doi: 10.1183/13993003.01209-2020. Print 2021 Apr. PMID 33033149
- [Derived] Tommola M, Won HK, Ilmarinen P, Jung H, Tuomisto LE, Lehtimaki L, Niemela O, Kim TB, Kankaanranta H. Relationship between age and bronchodilator response at diagnosis in adult-onset asthma. Respir Res. 2020 Jul 13;21(1):179. doi: 10.1186/s12931-020-01441-w. PMID 32660470
- [Derived] Ilmarinen P, Juboori H, Tuomisto LE, Niemela O, Sintonen H, Kankaanranta H. Effect of asthma control on general health-related quality of life in patients diagnosed with adult-onset asthma. Sci Rep. 2019 Nov 6;9(1):16107. doi: 10.1038/s41598-019-52361-9. PMID 31695074
- [Derived] Tommola M, Ilmarinen P, Tuomisto LE, Lehtimaki L, Niemela O, Nieminen P, Kankaanranta H. Cumulative effect of smoking on disease burden and multimorbidity in adult-onset asthma. Eur Respir J. 2019 Sep 5;54(3):1801580. doi: 10.1183/13993003.01580-2018. Print 2019 Sep. No abstract available. PMID 31048351